CLINICAL TRIAL: NCT06091592
Title: Serum autotaxın Level ın Colorectal Cancer
Brief Title: The dıagnostıc Value of Serum autotaxın Level ın Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, İsmail Oskay Kaya, PROFESSOR, Diskapi Yildirim Beyazit Education and Research Hospital
Other Study IDs: DYB-GC-AB-01
Record Dates: First submitted 2023-10-14; First posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Colo-rectal Cancer
Keywords: Colorectal cancer; autotaxın; biomarker
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — 5-10 ml of venous blood samples were taken from patients and healthy volunteers using blood collection tubes without anticoagulants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient ( cancer): . The colorectal cancer patient group included clinical stage 1-3 patients of both sexes. Patients with metastatic disease, those who received neoadjuvant therapy, those who received systemic chemoradiotherapy, those who had any known systemic inflammatory or autoimmune disease, those with another concurrent malignancy, and those who had been previously diagnosed and treated for another malignancy were excluded from the study.
  Interventions: Other: Serum autotaxın levels
- Control (healthy volunteer): The control group included healthy volunteers who had undergone screening colonoscopy within the last month, had no pathology, had not been diagnosed with any malignant disease before, had no known systemic inflammatory or autoimmune disease, and had not been diagnosed with inflammatory bowel disease.
  Interventions: Other: Serum autotaxın levels

INTERVENTIONS:
Other: Serum autotaxın levels — Autotaxin molecule is a nucleotide pyrophosphatase/phosphodiesterase enzyme.

SUMMARY:
Colorectal cancer is one of the most common causes of cancer-related death. Early diagnosis is extremely important in terms of treatment and mortality. In this study, we investigated the diagnostic value of serum autotaxin levels in colorectal cancer.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the third most common type of cancer worldwide. Among the causes of death due to cancer; it is the second most common among both genders with a rate of 9.2% after lung cancer . Early detection of the disease is important for survival. National screening programs attempt to detect this disease at an early stage.

Autotaxin (ATX) molecule is a member of the nucleotide pyrophosphatase/phosphodiesterase enzyme family (ENNP), It is secreted at 125 kDa, has lysophospholipase D activity in the lysophosphatidic acid (LPA) pathway, and is located at the 24th locus of the long arm of the 8th chromosome. This is also called ENPP2. It was discovered to be an autocrine motility-stimulating factor released by human melanoma A-2058 cells . Lysophosphatidic acid (LPA) is a lipid signalling molecule located in the cell membrane. LPA functions as an autocrine/paracrine messenger through at least six G protein-coupled receptors (GPCR) known as LPA 1-6. It plays physiologically important roles in various cellular processes, including wound healing, differentiation, cell proliferation, and migration. The role of ATX in the bioactivity of LPA is correlated with the lysophosphatidyl-D (lysoPLD) activity of ATX. ATX molecule; With this enzyme activity, it plays a fundamental role in the conversion of lysophosphatidylcholine to lysophosphatidic acid . Many studies have demonstrated the biological effects of the autotaxin-lysophosphatidic acid (ATX-LPA) signalling pathway in cancer. In vitro and in vivo studies have shown that increased ATX-LPA signalling contributes to cancer initiation and progression. Current evidence supports the role of the ATX-LPA signalling pathway in the proliferation, invasion, adhesion, and angiogenesis of cells, and is effective in cancer development and metastasis. Increased ATX expression has been reported in various cancers, such as glioblastoma, hepatocellular and thyroid carcinomas, breast, pancreatic, colon, and hematological cancers .

The ATX molecule has the feature of being a molecule that will be effective in the future, not only in the diagnosis of cancer, but also in the treatment process and to be studied extensively. in this study, we aimed to examine the diagnostic and biological behaviour relationship between serum ATX levels and colorectal cancer and to determine the cut-off value for serum ATX levels in colorectal cancer.

Serum ATX levels were compared between the patient and control groups. ATX levels were analysed in subgroups formed according to the demographic, clinical, pathological, and laboratory characteristics of the patient group.

ELIGIBILITY:
Inclusion Criteria:

* stage 1-3 colorectal cancer
* control group included healthy volunteers who had undergone screening colonoscopy within the last month , had no pathology,

Exclusion Criteria:

* metastatic disease,
* received neoadjuvant therapy
* received systemic chemoradiotherapy
* had any known systemic inflammatory or autoimmune disease
* had a with another concurrent malignancy
* had been previously diagnosed and treated for another malignancy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The colorectal cancer patient group included clinical stage 1-3 patients of both sexes. Patients with metastatic disease, those who received neoadjuvant therapy, those who received systemic chemoradiotherapy, those who had any known systemic inflammatory or autoimmune disease, those with another concurrent malignancy, and those who had been previously diagnosed and treated for another malignancy were excluded from the study. The control group included healthy volunteers who had undergone screening colonoscopy within the last month, had no pathology, had not been diagnosed with any malignant disease before, had no known systemic inflammatory or autoimmune disease, and had not been diagnosed with inflammatory bowel disease.
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2021-11-20 (Actual); Study Completion 2021-12-25 (Actual)

PRIMARY OUTCOMES:
Serum autotaxın level | one years
  The value measured by the Elisa method in blood samples taken from patients and healthy volunteers.

SECONDARY OUTCOMES:
Tumor location | one years
  It describes where this tumor is located in the colon in the patient group.
TNM stages | one years
  It describes the pathological staging of colorectal cancer patients.according to American Joint Committee on Cancer (AJCC) TNM system.
tumor differentiation grade | one years
  According to histopathological results, it is divided into three classes: well moderately and poor.

CONTACTS AND LOCATIONS:
Overall Officials: ismail o kaya, Principal Investigator — Dışkapı Yıldırım Beyazıt training and research hospital
Locations (1):
- Dışkapı Yıldırım Beyazıt training and research hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No